CLINICAL TRIAL: NCT00701844
Title: Sharing Our Strength: A Research Study for Bone Marrow/Stem Cell Transplant Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GCO #06-0391 (2); RSGPB-07-285-01-CPPB (Other: American Cancer Society)
Record Dates: First submitted 2008-06-04; First posted 2008-06-19 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2013-05

CONDITIONS: Leukemia; Acute Leukemia; Acute Lymphocytic Leukemia; Multiple Myeloma; Hematological Cancers; Psychological Distress
Keywords: Aplastic Anemia; Lymphatic Diseases; Leukemia; Leukemia, Lymphoid; Immunoproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia; Quality of Life; Lymphoproliferative Disorders; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma; Anemia, Aplastic; Lymphatic Diseases; Leukemia, Lymphoid; Immunoproliferative Disorders; Anemia; Lymphoproliferative Disorders; Lymphoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental Writing Type 1 (Experimental)
  Interventions: Behavioral: Writing A (Experimental informative writing)
- Experimental Writing type 2 (Experimental)
  Interventions: Behavioral: Writing B (Experimental noninformative writing)
- Control writing type 1 (Active Comparator)
  Interventions: Behavioral: Writing C (Control informative writing)
- Control writing type 2 (Placebo Comparator)
  Interventions: Behavioral: Writing D (Control noninformative writing)

INTERVENTIONS:
Behavioral: Writing A (Experimental informative writing) — Experimental informative writing
  Arms: Experimental Writing Type 1
Behavioral: Writing B (Experimental noninformative writing) — Experimental noninformative writing
  Arms: Experimental Writing type 2
Behavioral: Writing C (Control informative writing) — Control informative writing
  Arms: Control writing type 1
Behavioral: Writing D (Control noninformative writing) — Control noninformative writing
  Arms: Control writing type 2

SUMMARY:
The Sharing Our Strength study is being conducted to help us understand people's experiences with hematopoietic stem cell transplantation and to test a new program designed to help people recover physically and emotionally after transplant.

DETAILED DESCRIPTION:
This is a study for survivors of hematopoietic stem cell transplantation (also known as bone marrow transplant), which is an intensive medical treatment for cancers such as leukemia, lymphoma, and multiple myeloma as well as other diseases. Because it is a physically and emotionally demanding treatment, many people report having ongoing physical and emotional difficulties after having a transplant. The Sharing Our Strength study is being conducted to help us understand people's transplant experiences and to test a new program designed to help them recover physically and emotionally after transplant. All parts of the study are completed by mail and telephone. Participants will receive compensation for their time.

ELIGIBILITY:
Inclusion Criteria:

* Be a transplant survivor who is 9 months to 3 years beyond transplant and not currently relapsed. and not currently relapsed
* Be at least 18 years old now (and at least 16 when they had their transplant)
* Speak English
* Have telephone service

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2007-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Psychological Adjustment | At screening, baseline and 3 months following intervention

SECONDARY OUTCOMES:
Quality of Life | At screening, baseline and 3 months following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rini, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina